CLINICAL TRIAL: NCT02561000
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety of PZ-128 in Subjects Undergoing Non-Emergent Percutaneous Coronary Intervention- Thrombin Receptor Inhibitory Pepducin in PCI (TRIP-PCI)
Brief Title: Safety of PZ-128 in Subjects Undergoing Non-Emergent Percutaneous Coronary Intervention
Acronym: TRIP-PCI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); RTI International (Other); Inova Fairfax Hospital (Other); University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TMC-PZ128-02; P50HL110789 (NIH)
Record Dates: First submitted 2015-09-24; First posted 2015-09-25 (Estimated); Results first posted 2021-03-09 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2021-02

CONDITIONS: Arterial Occlusive Diseases; Coronary Artery Disease; Coronary Disease; Arteriosclerosis; Heart Diseases; Myocardial Ischemia; Vascular Diseases; Acute Coronary Syndrome
Keywords: Platelets; Platelet Aggregation Inhibitors; Protease-Activated Receptor 1; Hemorrhage
MeSH Terms: conditions — Arterial Occlusive Diseases; Coronary Artery Disease; Coronary Disease; Arteriosclerosis; Heart Diseases; Myocardial Ischemia; Vascular Diseases; Acute Coronary Syndrome; Hemorrhage | interventions — PZ-128 peptide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PZ-128 0.3 mg/kg (Experimental): PZ-128, 0.3 mg/kg, in 250 cc 5% dextrose, single dose, 2-hour intravenous infusion
  Interventions: Drug: PZ-128
- PZ-128 0.5 mg/kg (Experimental): PZ-128, 0.5 mg/kg, in 250 cc 5% dextrose, single dose, 2-hour intravenous infusion
  Interventions: Drug: PZ-128
- Placebo (Placebo Comparator): Placebo, in 250 cc 5% dextrose, single dose, 2-hour intravenous infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PZ-128
  Arms: PZ-128 0.3 mg/kg; PZ-128 0.5 mg/kg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The object of the study is to determine whether different doses of PZ-128, when added to standard medical care in persons undergoing cardiac catheterization/percutaneous coronary intervention, will increase the risk of bleeding.

A secondary objective is to determine whether patients treated with PZ-128 have fewer cardiac events such as heart attack, bypass surgery or stroke compared with those persons treated with the standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is at least 18 years of age and may be of either sex/gender and of any race and ethnicity.
2. The subject is scheduled to undergo non-emergent PCI or non-emergent cardiac catheterization with the intention of performing PCI. The following classifications of the urgency of the procedure at the time the operator decides to perform it will be used for randomization stratification:

   * Elective: The cardiac catheterization procedure ± PCI can be performed on an outpatient basis or during a subsequent hospitalization without significant risk of MI or death. For stable inpatients, this is a procedure that is performed during the hospitalization for convenience and ease of scheduling only and not because the subject's clinical situation demands that the procedure be performed prior to discharge.

   OR
   * Urgent: The cardiac catheterization ± PCI procedure should be performed on an inpatient basis and before discharge because of significant concerns about the risk of myocardial ischemia, MI and/or death. For subjects who are outpatients or in the emergency department at the time that the cardiac catheterization is requested, this is a procedure that would warrant hospital admission based on clinical presentation.
3. There is no anticipation that the subject would require treatment with a GP IIb/IIIa inhibitor prior to the initiation of the cardiac catheterization ± PCI procedure if the subject were not a participant in the current research study, and no anticipation of use during the procedure.
4. The subject is willing and able to give appropriate informed consent and complete all study-related procedures, and able to adhere to dosing and visit schedules (i.e., subject signs an approved informed consent document(s) and provides HIPAA authorization);
5. The subject will undergo all of the pre-enrollment parameters according to the study protocol prior to randomization and have them completed within 14 days prior to the scheduled cardiac catheterization ± PCI procedure and study drug administration.
6. Women of childbearing potential (all postmenarchal women who are <1 year menopausal or who have not had surgical sterilization or a hysterectomy are considered to be women of child-bearing potential) must agree to use a medically accepted method of contraception from the time written informed consent is given up until 90 days following the study drug administration.

Subject Exclusion Criteria:

The subject will be excluded from entry if any of the criteria listed below are met:

(General Exclusions)

1. Subject is pregnant, intends to become pregnant or is breast-feeding (all women of child-bearing potential must have a negative pregnancy test result confirmed prior to randomization and it must be repeated to be within 24 hours prior to the study drug administration if necessary).
2. Any of the following allergy history(s):

   * History of an allergic reaction* or contraindication to any of the following protocol-directed drugs: aspirin, heparin, P2Y12 inhibitor (clopidogrel, prasugrel, ticagrelor), antihistamines (benadryl, famotidine); or
   * History of an allergic reaction* to contrast media; or
   * History of an allergic reaction* to a drug which required emergency medical treatment;
   * History of an allergic reaction* to a Hymenoptera sting which currently necessitates the subject to carry an EpiPen/injector or the subject has been prescribed one to treat an allergic reaction to a sting.

     * An allergic (anaphylactic) reaction is characterized by an adverse local or general response from exposure to an allergen involving skin/mucosal tissue manifestations (hives, pruritus, flushing, angioedema), and/or respiratory compromise (dyspnea, wheeze-bronchospasm, stridor, reduced peak expiratory flow, hypoxemia), and/or hemodynamic effects (hypo/hypertension, hypotonia, syncope).
3. Participation in another research study of investigational therapy (drug or device) within the past 30 days prior to randomization or planned use of other investigational therapy(s) during this research study (until 90 days following the study drug administration).
4. Subject is part of the study staff personnel directly involved with this trial, or is a family member of the study staff (clinical site or sponsor).
5. Prior enrollment (randomization) in this research study.
6. Any condition which could interfere with, or the treatment for which might interfere with, the conduct of the research study or which would, in the opinion of the investigator, unacceptably increase the subject's risk by participating in the research study. This would include, but is not limited to alcoholism, drug dependency or abuse, psychiatric disease, epilepsy or any unexplained blackouts.

   (Exclusionary Prior/Concomitant Conditions)
7. Evidence of an ST-segment elevation myocardial infarction (STEMI) on presentation or during current hospitalization or a history of STEMI within the past 30 days prior to randomization.
8. Subject is scheduled to undergo PCI for known unprotected left main coronary artery (LMCA) disease (i.e., left main stenosis ≥50% not protected by at least 1 patent bypass graft).
9. Any history of a prior stroke (hemorrhagic or ischemic) or transient ischemic attack (TIA) of any etiology.
10. Cardiogenic or any type of shock on presentation or during current hospitalization (i.e., systolic blood pressure <90 mm Hg requiring vasopressor or hemodynamic support).
11. History of heparin-induced thrombocytopenia (HIT).
12. Any active bleeding within the past 30 days prior to randomization.
13. Any condition or personal belief (e.g., Jehovah's Witness) which would interfere with the subject's ability or willingness to undergo a blood transfusion.
14. Any of the following conditions associated with increased risk of bleeding:

    1. history of intracranial, intraocular, spinal, retroperitoneal or atraumatic intra- articular bleeding;
    2. gastrointestinal bleeding within the past 30 days prior to randomization;
    3. gastric or duodenal ulcer disease verified by endoscopy or barium meal contrast technique within the past 6 months prior to randomization;
    4. history of bleeding disorder or diathesis;
    5. major surgical procedure or trauma within the past 60 days prior to randomization or a planned surgical procedure to take place within 30 days following the study drug administration;
    6. history or suspicion of intracranial neoplasm, arteriovenous malformation, or aneurysm; or
    7. clinical finding(s) in the judgment of the investigator that poses an increased risk of bleeding.
15. Sustained severe hypertension: systolic blood pressure >185 mm Hg or diastolic blood pressure >105 mm Hg with or without anti-hypertensive treatment (as demonstrated by repeated BP measurements >185/105 mm Hg including the final BP measurement before randomization).
16. Hypotension: systolic blood pressure <95 mm Hg (as demonstrated by repeated systolic BP measurements <95 mm Hg including the final systolic BP measurement prior to randomization).
17. Known active hepatobiliary disease, or known unexplained persistent increase in serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) activity to ≥2.5 times the upper limit of the reference range within the past 30 days prior to randomization.
18. Hemoglobin <10 g/dL or hematocrit <30%.
19. Platelet count <75,000/mm3.
20. Stage 4-5 Chronic Kidney Disease (National Kidney Foundation) or on dialysis.
21. Active sepsis or suspected sepsis.
22. Body weight <60 kg or >175 kg.
23. Current evidence of invasive cancer (persistent disease excluding basal cell carcinoma of the skin) or treatment for invasive cancer within the past 6 months prior to randomization.
24. Left ventricular ejection fraction <25% if known (any imaging technique) or New York Heart Association (NYHA) Class IV congestive heart failure.

    (Exclusionary Prior/Concomitant/Anticipated Medication/Therapy)
25. Coronary interventional procedure of any kind within the past 30 days prior to randomization.
26. Anticipated subsequent staged multi-vessel PCI within 30 days following the study drug administration.
27. History of treatment with any parenteral GP IIb/IIIa inhibitor (GPI) within the past 30 days prior to randomization. (As stated in the Inclusion section, the planned treatment with a GPI prior to initiation of the cardiac catheterization ± PCI is not allowed; however, GPI for thrombotic bailout may be used during the PCI at the investigator's discretion).
28. Concurrent or anticipated treatment with a parenteral direct thrombin inhibitor (e.g., bivalirudin) for the cardiac catheterization ± PCI procedure.
29. History of treatment with another PAR1 inhibitor within the past 60 days prior to randomization or the concurrent/anticipated use after randomization up until 30 days following the study drug administration.
30. History of treatment with another IV anti-platelet drug within 30 days prior to randomization or the concurrent/anticipated use after randomization up until 30 days following the study drug administration.
31. Any of the following anticoagulant or thrombolytic/fibrinolytic treatment(s):

    * History of treatment with warfarin within 5 days prior to randomization or the concurrent/anticipated use after randomization up until 2 days following the study drug administration; or
    * History of treatment with oral Factor Xa or direct thrombin inhibitors within 2 days prior to randomization or the concurrent/anticipated use after randomization up until 2 days following the study drug administration; or
    * History of treatment with thrombolytic/fibrinolytic agents within 7 days prior to randomization or the concurrent/anticipated use of any of those agents after randomization up until 30 days following the study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-05-27 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Athan Kuliopulos, MD, PhD, Study Director — Tufts Medical Center
Locations (3):
- United States (3):
  - Tufts Medical Center, Boston, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Inova Heart and Vascular Institute, Inova Fairfax Hospital, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gurbel PA, Bliden KP, Turner SE, Tantry US, Gesheff MG, Barr TP, Covic L, Kuliopulos A. Cell-Penetrating Pepducin Therapy Targeting PAR1 in Subjects With Coronary Artery Disease. Arterioscler Thromb Vasc Biol. 2016 Jan;36(1):189-97. doi: 10.1161/ATVBAHA.115.306777. PMID 26681756
- [Result] Rana R, Huang T, Koukos G, Fletcher EK, Turner SE, Shearer A, Gurbel PA, Rade JJ, Kimmelstiel CD, Bliden KP, Covic L, Kuliopulos A. Noncanonical Matrix Metalloprotease 1-Protease-Activated Receptor 1 Signaling Drives Progression of Atherosclerosis. Arterioscler Thromb Vasc Biol. 2018 Jun;38(6):1368-1380. doi: 10.1161/ATVBAHA.118.310967. Epub 2018 Apr 5. PMID 29622563
- [Result] Kuliopulos A, Gurbel PA, Rade JJ, Kimmelstiel CD, Turner SE, Bliden KP, Fletcher EK, Cox DH, Covic L; TRIP-PCI Investigators. PAR1 (Protease-Activated Receptor 1) Pepducin Therapy Targeting Myocardial Necrosis in Coronary Artery Disease and Acute Coronary Syndrome Patients Undergoing Cardiac Catheterization: A Randomized, Placebo-Controlled, Phase 2 Study. Arterioscler Thromb Vasc Biol. 2020 Dec;40(12):2990-3003. doi: 10.1161/ATVBAHA.120.315168. Epub 2020 Oct 8. PMID 33028101
- [Derived] Fletcher EK, Wang Y, Flynn LK, Turner SE, Rade JJ, Kimmelstiel CD, Gurbel PA, Bliden KP, Covic L, Kuliopulos A. Deficiency of MMP1a (Matrix Metalloprotease 1a) Collagenase Suppresses Development of Atherosclerosis in Mice: Translational Implications for Human Coronary Artery Disease. Arterioscler Thromb Vasc Biol. 2021 May 5;41(5):e265-e279. doi: 10.1161/ATVBAHA.120.315837. Epub 2021 Mar 25. PMID 33761760

RESULTS

PARTICIPANT FLOW:
Recruitment Details: NCT02561000: Study TMC-PZ128-02 (TRIP-PCI Trial) was conducted at 3 centers in the U.S. between 27 May 2016 and 25 May 2018. A total of 3056 patients were screened for study and 100 patients were randomly assigned to treatment.
Pre-assignment Details: Of the 3056 patients pre-screened for study, 2956 patients were pre-screening failures, and 100 patients were randomly assigned to treatment. Of the 100 patients, 3 never received study drug (2 withdrew following randomization and 1 experienced an adverse event pre-dose), leaving 97 patients valid for the primary safety analysis. All randomized patients with at least 1 follow-up assessment (98 patients) were included in the intent-to-treat (ITT) analysis set for secondary efficacy analyses.
Groups:
- Placebo: Placebo, in 250 cc 5% dextrose, single dose, 2-hour intravenous infusion
  Placebo
- PZ-128 0.3 mg/kg: PZ-128, 0.3 mg/kg, in 250 cc 5% dextrose, single dose, 2-hour intravenous infusion
  PZ-128
- PZ-128 0.5 mg/kg: PZ-128, 0.5 mg/kg, in 250 cc 5% dextrose, single dose, 2-hour intravenous infusion
  PZ-128
Period: Overall Study
Arm/Group | Placebo | PZ-128 0.3 mg/kg | PZ-128 0.5 mg/kg
Started (Randomization) | 34 | 35 | 31
Safety Population (The Safety population included randomized participants who received any amount of the study drug dose of the double-blind IP infusion (summarized and analyzed as treated).) | 35 (Includes 1 additional patient who was assigned PZ-128 0.3 mg/kg but received placebo in error (evaluated as placebo for primary safety outcome and adverse events).) | 31 (Excludes 4 patients who did not receive the study drug as allocated: 1 patient received placebo in error and was evaluated as placebo for primary safety outcome and adverse events; 2 patients withdrew full consent immediately after randomization prior to receiving any study drug; and 1 patient had an adverse event shortly after randomization prior to receiving any study drug.) | 31
Intent-to-Treat (ITT) Population at 30 Days (The Intent-to-treat (ITT) population included all randomized participants, regardless of study drug intake, who underwent at least 1 follow-up assessment within 30 days after study drug dosing.) | 34 | 33 (Excludes 2 patients who withdrew full consent immediately after randomization.) | 31
Intent-to-Treat (ITT) Population at 90 Days (The Intent-to-treat (ITT) population included all randomized participants, regardless of study drug intake, who underwent at least 1 follow-up assessment after 30 days up until 90 days after study drug dosing.) | 33 (Excludes 1 patient who withdrew consent for follow-up 21 days after study drug dosing.) | 31 (Excludes 4 patients: 2 patients withdrew full consent immediately after randomization; 1 patient followed only for 30 day ITT outcome (did not receive any study drug due to adverse event post randomization); and 1 patient withdrew consent for follow-up 7 days after study drug dosing.) | 31
Completed (Completion of the 90-day follow-up time point after study drug dosing.) | 32 | 31 | 31
Not Completed | 2 | 4 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 0
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PZ-128 0.3 mg/kg | PZ-128 0.5 mg/kg | Total
Number analyzed (Participants) | 34 | 35 | 31 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (12.1) | 62.4 (11.0) | 63.2 (8.6) | 61.5 (10.8)
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 13 | 14 | 47
  >=65 years | 10 | 17 | 14 | 41
  >=75 years | 4 | 5 | 3 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 7 | 16
  Male | 27 | 33 | 24 | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 3
  Not Hispanic or Latino | 32 | 35 | 30 | 97
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 1 | 2 | 0 | 3
  White | 30 | 29 | 30 | 89
  More than one race | 1 | 3 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 34 | 35 | 31 | 100

OUTCOME MEASURES:

1. Primary Outcome: First Occurrence of Major Plus Minor Thrombolysis in Myocardial Infarction (TIMI) Bleeding Events; Number/Percentage of Observed Participants With Outcome Measure Events During the Study (Primary Safety)
Description: All suspected bleeding events positively adjudicated by CEC in a blinded fashion, were used in the reporting of the number/percentage of observed participants with a first occurrence of a TIMI major or minor bleeding event.
Time Frame: From initiation of study drug up to 30 days following study drug
Population: The Safety population included randomized participants who received any amount of the study drug dose of the double-blind IP infusion (summarized and analyzed as treated). Four patients assigned to PZ-128 0.3 mg/kg did not receive randomized treatment allocation: 1 patient received placebo in error and was evaluated as placebo for primary safety outcome and adverse events; 2 patients withdrew consent right after randomization; and 1 patient had an adverse event prior to receiving any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PZ-128 0.3 mg/kg | PZ-128 0.5 mg/kg
Number analyzed (Participants) | 35 | 31 | 31
Participants | 0 | 1 | 0

2. Secondary Outcome: First Occurrence of Major Adverse Cardiovascular Event (MACE); Number/Percentage of Observed Participants With Outcome Measure Events During the Study (Secondary Efficacy)
Description: All suspected MACE events positively adjudicated by Clinical Events Committee (CEC) in a blinded fashion, were used in the reporting of the number/percentage of observed participants with a first occurrence of the composite cardiovascular (CV) outcome measure comprised of CV death, non-fatal Myocardial Infarction (MI), non-fatal stroke (ischemic, hemorrhagic or unknown), recurrent ischemia requiring hospitalization, or urgent coronary revascularization. The number/percentage of observed participants with outcome measure events during the study were reported.
Time Frame: From randomization up to 30 days following study drug
Population: The Intent-to-treat (ITT) population included all randomized participants, regardless of study drug intake, who underwent at least 1 follow-up assessment within 30 days after study drug dosing. Two patients (PZ-128 0.3 mg/kg) could not be evaluated for the 30-day outcome due to complete study withdrawal shortly after randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PZ-128 0.3 mg/kg | PZ-128 0.5 mg/kg
Number analyzed (Participants) | 34 | 33 | 31
Participants | 2 | 0 | 0

3. Secondary Outcome: First Occurrence of Major Adverse Cardiovascular Event (MACE); Number/Percentage of Observed Participants With Outcome Measure Events During the Study (Secondary Efficacy)
Description: All suspected MACE events positively adjudicated by Clinical Events Committee (CEC) in a blinded fashion, were used in the reporting of the number/percentage of observed participants with a first occurrence of the composite cardiovascular (CV) outcome measure comprised of CV death, non-fatal Myocardial Infarction (MI), non-fatal stroke (ischemic, hemorrhagic or unknown), recurrent ischemia requiring hospitalization, or urgent coronary revascularization.
Time Frame: From randomization up to 90 days following study drug
Population: The Intent-to-treat (ITT) population included all randomized participants, regardless of study drug intake, who underwent at least 1 follow-up assessment after 30 days up until 90 days after study drug dosing. 5 patients could not be evaluated for the 90-day outcome: 1 placebo withdrew at 21 d; 2 PZ-128 0.3 mg/kg withdrew post randomization; 1 PZ-128 0.3 mg/kg withdrew at 7 d; and 1 PZ-128 0.3 mg/kg patient was followed only for 30 d ITT outcome (no study drug due to AE post randomization).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PZ-128 0.3 mg/kg | PZ-128 0.5 mg/kg
Number analyzed (Participants) | 33 | 31 | 31
Participants | 2 | 0 | 1

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs), including Serious Adverse Events (SAEs), were collected from signature of the informed consent form until 30 days post study drug regardless of relationship to Investigational Product (IP).
Description: Reported AEs are treatment-emergent AEs that is AEs that developed/worsened during the 'treatment-emergent period' (the time from the study drug dosing up to 30 days post dose). Adverse Events do not include Study Endpoint Events. The Safety population included randomized participants who received any amount of the study drug dose of the double-blind IP infusion (summarized and analyzed as treated)- See Safety Population Milestone in Participant Flow Overview.
Arm/Group | Placebo | PZ-128 0.3 mg/kg | PZ-128 0.5 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 1/35 | 5/31 | 2/31
Other Adverse Events (participants affected / at risk) | 6/35 | 8/31 | 16/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=35) | PZ-128 0.3 mg/kg (N=31) | PZ-128 0.5 mg/kg (N=31)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Unrelated to study drug
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) — Unrelated to study drug
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Unrelated to study drug. Underwent index procedure cardiac catheterization and study drug for non-ST-elevation myocardial infarction. Patient has past medical history of atrial fibrillation and cardiomyopathy/left ventricular systolic dysfunction.
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) — Unrelated to study drug
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — Unrelated to study drug. Underwent index procedure cardiac catheterization + PCI and study drug for unstable angina. Patient has past medical history of heart failure with reduced left ventricular ejection fraction.
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) — Related to study drug
Aortic Valve Disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Unrelated to study drug. Underwent index procedure cardiac catheterization + PCI and study drug for non-ST-elevation myocardial infarction. Patient has past medical history of aortic valve disease.
Fluid Overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) — Unrelated to study drug. Underwent index procedure cardiac catheterization + PCI and study drug for non-ST-elevation myocardial infarction. Patient has past medical history of heart failure.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=35) | PZ-128 0.3 mg/kg (N=31) | PZ-128 0.5 mg/kg (N=31)
Atrial Fibrillation (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Hypoesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Paresthesia Oral (Nervous system disorders) | 0 (0) | 5 (5) | 6 (6)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 5 (5)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-04): https://cdn.clinicaltrials.gov/large-docs/00/NCT02561000/Prot_SAP_000.pdf